CLINICAL TRIAL: NCT03127462
Title: Efficiency of a Nurse-led Individualized Educational Intervention in Newly Referred Patients With Psoriasis. A Pragmatic Controlled Study.
Brief Title: A Nurse-led Individualized Educational Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lina R. Khoury (Other)
Responsible Party: Sponsor-Investigator, Lina R. Khoury, Ph.D student, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UA-1502
Record Dates: First submitted 2017-03-30; First posted 2017-04-25 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: In the first phase of the study 30 patients will receive standard treatment (control group) and in the following phase 30 patients will receive the individualized conversational/educational intervention (intervention group).The rationale for using a historical control group instead of a randomised control group is that it in"real-life setting" is unpractical to realize a communicative intervention, because clinicians unintentional can intervene against the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Education (Experimental)
  Interventions: Behavioral: Nurse-led educational intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Nurse-led educational intervention — Patients in the intervention group will receive an individual face-to-face conversation with a duration of 45 min. All patients will have access to telephone counselling by their primary nurse when needed and able to arrange a new face-to-face conversation. After 4-6 weeks the face-to-face the nurse will of conversation reach out to the patient by phone to follow up on the earlier conversation. Three months after the face-to-face conversation the nurse will offer the patient a closing face-to-face conversation of 15 min at the same time where the patient has a doctor appointment at the department. Those who are in the control group will continue standard care and not receive any conversation and be used as the control group.
  Arms: Individualized Education

SUMMARY:
60 newly referred patients with psoriasis at the Department of Dermatology and Allergy, Herlev and Gentofte Hospital, Denmark will be consecutive included in the study. In the first phase of the study 30 patients will receive standard treatment (control group) and in the following phase 30 patients will receive the individualized conversational/educational intervention (intervention group).The rationale for using a historical control group instead of a randomised control group is that it in"real-life setting" is unpractical to realize a communicative intervention, because clinicians unintentional can intervene against the control group.

The first conversation will take place when the newly referred patient has initiated a new treatment. The rational for this is that the time of transition from private practice to the Department of Dermatology and Allergy is characterised by failed treatment, typically phototherapy or topical. This meaning that newly referred patients current needs is to get their psoriasis under control. When patients have initiated a medical treatment they will be more motivated and have better surplus to engage in the conversational/educational intervention.

Patients in the intervention group will receive an individual face-to-face conversation with a duration of 45 min. All patients will have access to telephone counselling by their primary nurse when needed and able to arrange a new face-to-face conversation. After 4-6 weeks the face-to-face the nurse will of conversation reach out to the patient by phone to follow up on the earlier conversation. Three months after the face-to-face conversation the nurse will offer the patient a closing face-to-face conversation of 15 min at the same time where the patient has a doctor appointment at the department. Those who are in the control group will continue standard care and not receive any conversation and be used as the control group.

The intervention will be provided by a team of specialized dermatological nurses who have received a formal training on patient-centred communication, Self-regulatory Model/Common Sense Model interviewing, the life with chronic disease and action plan support.

ELIGIBILITY:
Inclusion Criteria:

* Newly referred patients with psoriasis at the Department of Dermatology and Allergy, Herlev and Gentofte Hospital, 18 years or older and understand Danish.

Exclusion Criteria:

* Patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
The brief Illness Perception Questionnaire | Change from Baseline at 3 month follow-up
  Illness perception

SECONDARY OUTCOMES:
Dermatology Life Quality Index | Change from Baseline at 3 month follow-up
  Quality of life

OTHER OUTCOMES:
The Patient Assessment of Chronic Illness Care | Change from Baseline at 3 month follow-up
  Perception of Care
Hospital Anxiety and Depression Scale | Change from Baseline at 3 month follow-up
  Anxiety and depression
Body Image Scale | Change from Baseline at 3 month follow-up
  Body image
Understanding of psoriasis | Change from Baseline at 3 month follow-up
  Patients understanding of psoriasis by a self-developed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No